CLINICAL TRIAL: NCT07025811
Title: A Longitudinal, Open-label, Multi-center Study to Explore the Relationship Between Signs, Symptoms, Molecular and Imaging Biomarkers in Participants With Dry Eye Disease Following Anti-inflammatory Treatment
Brief Title: A Study to Explore Signs, Symptoms, and Biomarkers in Dry Eye Disease Participants Following Anti-inflammatory Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP45931
Record Dates: First submitted 2025-06-16; First posted 2025-06-18 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Masking Description: This is a partially masked study where health care professionals conducting the ocular assessments will be masked to treatment assignment but not to study eye assignment. However, other site personnel and participants will be unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vevye® (Experimental): Participants with evaporative dry eye (EDE), aqueous deficient dry eye (ADDE) and mixed dry eye will receive Vevye®, 1 milligrams per milliliter (mg/mL) as one drop into the affected eye(s), twice daily (BID) via topical ocular instillation for 12 weeks.
  Interventions: Drug: Vevye®
- Xiidra® (Experimental): Participants with EDE, ADDE, and mixed dry eye will receive Xiidra®, 50 mg/mL as one drop into the affected eye(s), BID via topical ocular instillation for 12 weeks.
  Interventions: Drug: Xiidra®
- Healthy Cohort (No Intervention): Healthy volunteers will be enrolled as a control group and will not receive any treatment.

INTERVENTIONS:
Drug: Vevye® — Participants will receive Vevye® (0.1% cyclosporine ophthalmic solution) as per the schedule described in the treatment arm.
  Other Names: Cyclosporine Ophthalmic Solution
  Arms: Vevye®
Drug: Xiidra® — Participants will receive Xiidra® (5% lifitegrast ophthalmic solution) as per the schedule described in the treatment arm.
  Other Names: Lifitegrast Ophthalmic Solution
  Arms: Xiidra®

SUMMARY:
This study aims to evaluate the performance of biomarkers and their responsiveness to standard-of-care treatments (Vevye® or Xiidra®), in participants with dry eye disease (DED) compared to healthy volunteers (control participants).

DETAILED DESCRIPTION:
This study aims to characterize longitudinal changes in signs, symptoms, molecular, and imaging markers of the ocular surface to investigate pathological mechanisms and biomarkers (BMs) of DED after treatment with either of two commercially approved therapeutics (Vevye® [cyclosporine ophthalmic solution], Xiidra® [liftegrast ophthalmic solution]).

ELIGIBILITY:
Inclusion Criteria:

A. Inclusion Criteria for Participants with DED:

* The participant reported dry eye-related ocular symptoms for at least 6 months before the screening visit
* The participant must have either used lubricant eye drops regularly OR had the desire to use lubricant eye drops in the past 3 months
* Participant must be classified as having moderate/severe DED
* The participant is deemed by the physician to require a prescription medication for DED (e.g., cyclosporin A or lifitegrast)

B. Inclusion Criteria for Healthy Volunteers:

- The participant does not have overt clinical signs of DED in either eye

Exclusion Criteria:

* Intraocular pressure (IOP) >21.00 millimeters of mercury (mmHg) in either eye
* Acute allergic conjunctivitis in either eye within 3 months prior to screening
* Use of contact lenses within 30 days prior to screening
* Punctal plugs within 3 months prior to screening or any history of punctal cauterization or occlusion by an approach different from punctal plugs
* Use of ocular anti-inflammatory agents or ocular immunosuppressive agents within 3 months prior to screening
* Any intraocular injections (e.g., intravitreal [IVT] anti-vascular endothelial growth factor [VEGF]) within 3 months prior to screening, or such injections planned for within the study period
* Any intraocular immunosuppressive implants within 12 months prior to screening
* Any history of isotretinoin use within 12 months prior to screening
* Uncontrolled ocular or systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Corneal Staining as Measured by Sodium Fluorescein | Up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Andover Eye Associates, Andover, Massachusetts
  - Oculus Research, Garner, North Carolina
  - Total Eyecare, P.A., Memphis, Tennessee
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing